CLINICAL TRIAL: NCT02628002
Title: Comparison of Anti-gravity Treadmill Exercise and Regadenoson Tc-99m Tetrofosmin Single-photon Emission Computed Tomography (SPECT) Myocardial Perfusion Imaging
Brief Title: Anti-gravity Treadmill Exercise in Stress Myocardial Perfusion Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Myron C. Gerson, professor emeritus of Cardiology, University of Cincinnati
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2014-5363
Record Dates: First submitted 2015-03-24; First posted 2015-12-11 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Coronary Artery Disease
Keywords: antigravity treadmill; bruce protocol; stress myocardial perfusion imaging; single photon emission computed tomography; cardiac catheterization; [E01.370.370.380.500]; [E01.370.370.380.250]; [E01.370.370.380.140]
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test arm (Experimental): The subjects randomized to the anti-gravity treadmill arm will be instructed on the safe use of the Alter-G treadmill by the study staff. After this instruction, subjects will be exercised on the Alter-G anti-gravity treadmill using the conventional Bruce protocol with unweighting to 75% of their body weight to reach target heart rate. If the subject is unable to reach the target heart rate, they will be further unweighted to 50% of their body weight to enable the subject to reach target heart rate on the Bruce protocol. If the subject is still unable to reach target heart rate with 50% unweighting, the patient's subsequent SPECT images will be excluded from use in the research comparison to control subject images.
  Interventions: Device: Antigravity treadmill (Alter-G)
- Control arm (Active Comparator): The control arm subjects will undergo the conventional treadmill/regadenoson pharmacological stress SPECT. Consistent with standard practice, these patients will perform adjunctive low-intensity walk on a conventional treadmill prior to regadenoson and Tc-99m injection if tolerated.
  Interventions: Device: Conventional treadmill/regadenoson

INTERVENTIONS:
Device: Antigravity treadmill (Alter-G) — Test arm subjects will exercise according to the Bruce protocol unweighted to 75% of their body weight with additional unweighting to 50% during the test if unable to reach target at 75% weight. Once these subjects have reached their target heart rate on the Bruce protocol, patients will receive the Tc-99m injection as per standard clinical protocol and maintain target heart rate for 1 minute following the injection.
  Arms: Test arm
Device: Conventional treadmill/regadenoson — Subjects randomized to the control arm will proceed with the clinical standard regadenoson pharmacological stress SPECT study with adjunctive low-intensity walk on conventional treadmill during regadenoson and Tc-99m injections if tolerated. If they are unable to tolerate any treadmill exercise, they will receive regadenoson and Tc-99m injections at rest. Study patients will have stable systemic blood pressure with readings equal to or greater than 90 mmHg systolic. Other inclusion and exclusion criteria are described in detail below.
  Arms: Control arm

SUMMARY:
This study will test the hypothesis that the anti-gravity treadmill can be safely used in stress nuclear myocardial perfusion imaging in patients unable to perform conventional treadmill exercise.

This will be foundational evidence on which to consider a larger clinical trial to show that the anti-gravity treadmill improves diagnostic specificity across all cardiovascular stress testing modalities including treadmill-alone, exercise stress echocardiogram, exercise SPECT as well as having implications for cardiac PET and MRI in the future.

DETAILED DESCRIPTION:
This randomized, single blind, controlled study will enroll up to 75 subjects presenting to the nuclear cardiology stress lab for a previously ordered SPECT study. Potential subjects will be identified by the study staff and stress lab staff prior to the stress portion of their study when the potential subject states an inability to exercise to target heart rate on the conventional treadmill prior to starting exercise. The study coordinator will then be contacted to obtain informed consent from the study subject. Subjects, after signing an informed consent document, will be enrolled and will complete the enrollment. If the subject qualifies for the study, they will then be randomized with a 2:1 ratio between the test and control arms using a preprinted randomization table.

Subjects randomized to the test arm will be instructed on the proper procedure for safely entering and exercising on the anti-gravity treadmill by the stress lab and research staff. Subjects will be provided a size-appropriate pair of neoprene shorts to be worn over their clothes. The shorts attach to the anti-gravity treadmill. These shorts will be cleaned following each patient use. Test arm subjects will exercise according to the Bruce protocol unweighted to 75% of their body weight with additional unweighting to 50% during the test if unable to reach target at 75% weight. Once these subjects have reached their target heart rate on the Bruce protocol, patients will receive the Tc-99m injection as per standard clinical protocol and maintain target heart rate for 1 minute following the injection. Patients will then be brought to walk speed for recovery.

Any subject in the test arm who is unable to reach target heart rate on the anti-gravity treadmill will be slowed to walk speed and receive regadenoson and Tc-99m injections while walking. They will be maintained at 75% unweighting while walking for these injections. Subjects unable to reach target on the anti-gravity treadmill will be included in the final data safety analysis but will be excluded from the test arm image analysis.

Subjects randomized to the control arm will proceed with the clinical standard regadenoson pharmacological stress SPECT study with adjunctive low-intensity walk on conventional treadmill during regadenoson and Tc-99m injections if tolerated. If they are unable to tolerate any treadmill exercise, they will receive regadenoson and Tc-99m injections at rest. Study patients will have stable systemic blood pressure with readings equal to or greater than 90 mmHg systolic. Other inclusion and exclusion criteria are described in detail below.

All images will be acquired by the standard clinical imaging protocol and processed by a trained nuclear medicine technologist. The imaging will then be analyzed and read by an experienced nuclear cardiologist who is blinded to whether patient is in the anti-gravity treadmill or control arm. The subsequent images and values will be confirmed by a separate and blinded experienced nuclear cardiologist. The uptake counts of isotope in the left ventricle versus the background counts will be recorded and compared between the test arm and the control arm.

ELIGIBILITY:
Inclusion Criteria:

1. Patients >18 years of age who are able to ambulate.
2. Women will either have a negative pregnancy test, be post-menopausal or have prior surgical infertility
3. Nuclear stress SPECT imaging test ordered as exercise SPECT or regadenoson SPECT.
4. If ordered for exercise SPECT, self-admission of inability to exercise on conventional treadmill. This typically includes subjects unable to exercise due to obesity, musculoskeletal disease, peripheral vascular disease, weakness or debilitation.
5. Patients that initially start conventional treadmill exercise protocol and have to stop due to exercise-limiting symptoms including musculoskeletal pain and fatigue.
6. Hemodynamically stable patients as defined by mean blood pressure (BP) >75 mm Hg and heart rate (HR) 60-120 beats per minute.

Exclusion Criteria:

1. Hemodynamically unstable patients as defined by resting mean BP <75 and HR <60 or >120.
2. Patients with acute coronary syndrome as defined by troponin elevation (>0.05) within the past 72 hours.
3. Patients at high clinical risk related to severe aortic stenosis, known exercise-induced ventricular tachycardia or fibrillation, or advanced (second-degree type II or third-degree) heart block.
4. Patients with left bundle branch block or paced cardiac rhythm (in whom exercise is associated with non-ischemic perfusion abnormalities).
5. Patients unable to provide consent or unable to cooperate.
6. Inability to physically enter onto the anti-gravity treadmill unit.
7. Pregnant women.
8. Patients with a contraindication to receive regadenoson (sinus node dysfunction, high-degree heart block, active wheezing/reactive airway disease).
9. At risk patient populations (prisoners or severely mentally handicapped).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Safely Reach Target Heart Rate on the Anti-Gravity Treadmill | 1 year
  Patients who are unable to perform conventional treadmill exercise will be exercised to target heart rate on the anti-gravity treadmill for stress nuclear myocardial perfusion imaging.

SECONDARY OUTCOMES:
Effect of Anti-Gravity Treadmill Exercise on Heart Rate | 1 year
  Heart rate associated with physiologic exercise on the anti-gravity treadmill measured in patients being evaluated with myocardial perfusion imaging.
Effect of Anti-Gravity Treadmill Exercise on Blood Pressure | 1 year
  Blood pressure associated with physiologic exercise on the anti-gravity treadmill measured in patients being evaluated with myocardial perfusion imaging.
Perfusion Imaging Quality After Anti-Gravity Treadmill Exercise | 1 year
  The quality of the resulting perfusion images will be compared following exercise on the conventional treadmill versus anti-gravity treadmill.

CONTACTS AND LOCATIONS:
Overall Officials: Myron Gerson, MD, Principal Investigator — University of Cincinnati; Patrick Daly, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No